CLINICAL TRIAL: NCT05167344
Title: Evaluation of the Healthy Relationships Program-Enhanced (HRP-E) for Vulnerable Youth
Acronym: HRP-E
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Western University, Canada (Other)
Responsible Party: Principal Investigator, Claire Crooks, Professor; Director, Centre for School Mental Health, Western University, Canada
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: WREM 120133
Record Dates: First submitted 2021-11-10; First posted 2021-12-22 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Adolescent Behavior; Dating Violence
Keywords: vulnerable youth; social-emotional functioning; dating violence; mental health
MeSH Terms: conditions — Adolescent Behavior; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Youth and facilitators participating in HRP-E program (intervention arm)
Masking Description: Due to the nature of the intervention, it is not possible to have blinded conditions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy Relationships Program-Enhanced (HRP-E) (Experimental): Youth participating in the HRP-E and facilitators delivering in the program
  Interventions: Behavioral: Healthy Relationships Program-Enhanced

INTERVENTIONS:
Behavioral: Healthy Relationships Program-Enhanced — The Healthy Relationships Program-Enhanced (HRP-E) is a small group mental health promotion and healthy relationship program designed for vulnerable, at-risk youth. It is a trauma-informed, 16-session manualized program.

SUMMARY:
Investigators will work with community partners to undertake an evaluation of the impact of the Healthy Relationships Program-Enhanced (HRP-E) for youth to build evidence on effective programming with diverse vulnerable youth populations in real-world contexts. Youth participants will complete four surveys before and after participating in the HRP-E program and an interview approximately 4 to 6 months after participating in the program. Program facilitators will also track session activities and youth participation throughout the program and are invited to participate in a survey after the program is complete.

DETAILED DESCRIPTION:
Study Background and Design:

Vulnerable youth disproportionately experience dating violence, trauma, abuse, and maltreatment. Vulnerable youth are defined as youth at risk of, or currently experiencing, harm or adversities due to social and environmental factors. Youth who have experienced violence, trauma, abuse, and maltreatment have a more difficult time developing healthy, stable relationships in adolescence and beyond. They also often become involved in community mental health care, welfare care, and the justice system. Vulnerable youth are in need of programming to provide education and skill-building in areas such as healthy relationships, mental health, and substance use. Many stakeholders, including university-based researchers and community partners, recommend integrating mental health interventions into settings where youths are already receiving essential services (e.g., schools, child welfare agencies).

The Healthy Relationships Program-Enhanced (HRP-E) fills a gap in mental health promotion and healthy relationship programming. It is a trauma-informed, 16-session manualized program designed to be facilitated in small group settings by educators or community professionals. The program's core components derive from the evidence-based, Canadian Fourth R program, a classroom-based, universal healthy relationships promotion and dating violence prevention curriculum (Crooks et al., 2011, 2015; Wolfe et al., 2009, 2012). The HRP-Enhanced program has been successfully implemented in various settings (e.g., schools, youth corrections). However, the impact of the program on vulnerable youth has not been extensively studied and needs to be further examined to under the effectiveness of this program across diverse settings (e.g., community mental health services, child welfare services, juvenile justice).

Investigators will work with our community partners to undertake a mixed-methods evaluation, including repeated measures time-series survey and follow-up interviews, to examine the impacts of the HRP-Enhanced Program to build evidence on what type of programming works with diverse vulnerable youth populations. Program facilitators will track session activities and youth participation throughout the program, and participate in a post-program implementation. Specifically, investigators will be able to determine the extent to which the HRP-E promotes positive mental health and well-being among vulnerable youth and identify changes in social-emotional assets and resilience, youth well-being, mental health, dating violence and help-seeking.

Participants:

Youth participating in HRP-E and program facilitators are eligible to participate in this study. Investigators will work with each community partner to identify 2 to 4 HRP-E groups they are delivering to be invited to participate in this research study (a total of 20 groups). Approximately 100-150 youth are expected to participate in this study, and approximately 10 to 20 facilitators. The number of youth and facilitators will be dependent on the number of HRP-Enhanced groups delivered and the total number of youth participating in the program.

Procedures:

Youth will be invited to participate in three research activities: a survey at four time-points, individual interviews, and providing consent for the use of program session tracking information collected by facilitators on their participation in the program for research purposes. (note: the session tracking data are collected routinely by facilitators, so it is the use of those data that participants are consenting to, not the collection).

The survey is administered at four time-points: i) two weeks to one month before they start the program (baseline); ii) at the start of the program (pre-intervention); iii) at the end of the program (post-intervention), and; iv) one month after the end of the program (follow-up). The survey asks questions about youths' mental health and well-being, who they might seek support from, dating and dating violence, bullying, and questions about their identities. The interview will take place approximately 4 to 6 months after the youth completes the program. The semi-structured interview asks youth about their experiences participating in the program and any skills they have learned and used.

The session tracking data includes youths' attendance, perceived engagement (as rated by the facilitator), and any trauma-related behaviours shown in group (as rated by facilitator). If youth consent to the sharing of those data, they will be de-identified by facilitators and shared with a unique participant identifier (ID) to facilitate merging of data across sources.

Facilitators implementing the HRP-E program will be invited to share their quality improvement data from their session tracking sheets for research purposes. They are also invited to complete an online implementation survey at the end of the HRP-Enhanced group to understand their experiences implementing the program with the recent HRP group they facilitated. The survey includes questions regarding group and facilitator characteristics, group format and logistics, virtual considerations, modifications, and program impact.

Planned Analyses:

Investigators will explore the baseline and pre-intervention data through bivariate analyses to investigate significant differences in outcomes and regression to the mean. If no significant differences, a new time 1 variable will be calculated using the mean of time 1 and time 2. Bivariate comparisons will be completed between pre-intervention and post-intervention outcomes, as well as pre-intervention and follow-up outcomes. Effect sizes will be calculated using Cohen's d. Analyses will also include general linear model (GLM) repeated measures to examine potential gender effects and/or time-by-gender interactions related to post-intervention outcomes. Finally, chi-square analyses will be conducted to determine whether systematic attrition occurred.

ELIGIBILITY:
Inclusion Criteria:

* Youth participating in the Healthy Relationships Program-Enhanced
* Facilitators delivering the Healthy Relationships Program-Enhanced
* A minimum of three youth participating as a group in the Healthy Relationships Program-Enhanced

Exclusion Criteria:

* Youth with low literacy or cognitive functions who may not be able to complete the self-report measures

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-04-14 (Actual); Primary Completion 2023-04-01 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
Positive social-emotional functioning | Change from baseline to one-month post program completion (up to 20 weeks)
  Measured by the Social-Emotional Assets and Resiliency Scales-Adolescent (SEARS-A) that assesses social-emotional assets of responsibility, self-regulation, social competence, and empathy. Participants respond to the 35 items on a 4-point Likert scale (0 = never, 1 = sometimes, 2 = often, 3 = always). The combined total score ranges from 0 to 105 with higher scores indicating greater social-emotional strengths.

SECONDARY OUTCOMES:
Dating Violence | Change from baseline to one-month post program completion (up to 20 weeks)
  Dating violence perpetration as measured by the Conflict in Adolescent Dating Relationships Inventory (short form). Participants respond to the 20 items on a 4-point Likert scale (0 = never, 1 = seldom, 2 = sometimes, 3 = often). The sum of the perpetrator and victimization items are calculated (10 items each). Scores range from 0 to 30 with higher scores indicating a higher incidence of abusive behaviour (perpetrator items) or victim of abuse (victimization items).
Help-seeking intentions | Change from baseline to one-month post program completion (up to 20 weeks)
  Self-reported intentions to seek help as measured by General Help-seeking Questionnaire. Participants indicate their likelihood to seek help for a personal or emotional problem from the people listed on a 4-point Likert scale (1= very unlikely, 2=unlikely, 3=likely, 4=very likely). A mean score is calculated on the items with the higher score indicating a higher likelihood to seek help for a problem.
Actual help-seeking | Change from baseline to one-month post program completion (up to 20 weeks)
  Actual help-seeking over the past 2 weeks as measured by the Actual Help Seeking Questionnaire. Participants check the people they have sought help from over a two-week period for a personal or emotional problem and then describe the type of problem. A score for the total number of people they sought help from is calculated and open-ended descriptions are coded for type of problem (e.g., mental health, relationships, school, etc.).
Positive mental health | Change from baseline to one-month post program completion (up to 20 weeks)
  Emotional well-being and aspects of psychological and social functioning that occur within the past month as measured by the Adolescent Mental Health Continuum-Short Form. Participants rate 14 items on a 6-point Likert scale from 0=Never to 5 = Every day. Scores range from 0 to 70 with higher scores indicating higher experience of positive mental health.
Emotional distress | Change from baseline to one-month post program completion (up to 20 weeks)
  Stress and depression items from modified Depression Anxiety Stress Scales (DASS-21). Participants rate the 14 stress and depression items on a 4-point Likert scale from 0=never to 3 = more than two times. Total scores are calculated for the stress and depression subscales with a range of 0 to 21 with higher scores indicating higher stress or depression.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Claire Croooks, PhD, Principal Investigator — Western University
Locations (1):
- Western University, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Andrews, N., Pepler, D., Motz, M. (2019). Research and evaluation with community-based projects: Approaches, considerations, and strategies. American Journal of Evaluation, 40(4), 548-561. https://doi.org/10.1177/1098214019835821
- [Background] Antle, B. F., Sullivan, D. J., Dryden, A., Karam, E. A., & Barbee, A. P. (2011). Healthy relationship education for dating violence prevention among high-risk youth. Children and Youth Services Review, 33(1), 173-179. doi:10.1016/j.childyouth.2010.08.031
- [Background] Crooks CV, Scott K, Ellis W, Wolfe DA. Impact of a universal school-based violence prevention program on violent delinquency: distinctive benefits for youth with maltreatment histories. Child Abuse Negl. 2011 Jun;35(6):393-400. doi: 10.1016/j.chiabu.2011.03.002. Epub 2011 Jun 8. PMID 21652072
- [Background] Crooks CV, Scott KL, Broll R, Zwarych S, Hughes R, Wolfe DA. Does an evidence-based healthy relationships program for 9th graders show similar effects for 7th and 8th graders? Results from 57 schools randomized to intervention. Health Educ Res. 2015 Jun;30(3):513-9. doi: 10.1093/her/cyv014. Epub 2015 Apr 2. PMID 25840436
- [Background] Smyth, P. (2017). Working with high-risk youth: A relationship-based practice framework. Routledge Academic. London: Routledge, https://doi.org/10.4324/9781315270043
- [Background] Wekerle C, Leung E, Wall AM, MacMillan H, Boyle M, Trocme N, Waechter R. The contribution of childhood emotional abuse to teen dating violence among child protective services-involved youth. Child Abuse Negl. 2009 Jan;33(1):45-58. doi: 10.1016/j.chiabu.2008.12.006. Epub 2009 Jan 22. PMID 19167066
- [Background] Wolfe DA, Crooks C, Jaffe P, Chiodo D, Hughes R, Ellis W, Stitt L, Donner A. A school-based program to prevent adolescent dating violence: a cluster randomized trial. Arch Pediatr Adolesc Med. 2009 Aug;163(8):692-9. doi: 10.1001/archpediatrics.2009.69. PMID 19652099
- [Background] Wolfe DA, Crooks CV, Chiodo D, Hughes R, Ellis W. Observations of adolescent peer resistance skills following a classroom-based healthy relationship program: a post-intervention comparison. Prev Sci. 2012 Apr;13(2):196-205. doi: 10.1007/s11121-011-0256-z. PMID 22057307